CLINICAL TRIAL: NCT06198140
Title: Effects of Myofascial Release With and Without Quick Icing on Tone, Range of Motion and Balance in Children With Cerebral Palsy
Brief Title: Effects of Myofascial Release in Cerebral Palsy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC/RCR&AHS/23/0750
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Myofascial Release; Range of motion; Quick icing
MeSH Terms: conditions — Cerebral Palsy | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Release and Quick icing (Experimental): Experimental group will receive myofascial release & quick icing.
  Interventions: Other: myofascial release and quick icing
- Myofascial Release (Active Comparator): In control group the individuals will receive only myofascial release on ankle planterflexors.
  Interventions: Other: myofascial release

INTERVENTIONS:
Other: myofascial release and quick icing — In experimental group the individuals will receive myofascial release and quick icing. Quick icing will be on ankle dorsiflexors by using ice pack in the target area. Quick icing will be applied for 10 minutes (time of application 10 seconds and a rest for 20 seconds). This treatment protocol will be 6 times/week for 4 weeks in the hospital setting. Mayofascial release will be given on the target ankle planterflexors. The subjects who will receive Myofascial Release will be positioned in prone with the treatment area exposed. The treatment will be applied by the therapist standing at the side of the patient. Then technique will be applied with different levels by following longitudinal movements according to subject's tolerance for duration of 3 minutes in each sitting. Patients will be given a rest time after each level in order to allow the tissue to soften. This treatment protocol will be 6 times/week for 4 weeks in the hospital setting.
  Arms: Myofascial Release and Quick icing
Other: myofascial release — In control group the individuals will receive only myofascial release on ankle planterflexors. The subjects who will receive Myofascial Release will be positioned in prone with the treatment area exposed. The treatment will be applied by the therapist standing at the side of the patient. Then technique will be applied with different levels by following longitudinal movements according to subject's tolerance for duration of 3 minutes in each sitting. Patients will be given a rest time after each level in order to allow the tissue to soften. This treatment protocol will be 6 times/week for 4 weeks in the hospital setting.
  Arms: Myofascial Release

SUMMARY:
Cerebral palsy (CP) is a common disorder which leads to physical disability in children throughout life and begins in early childhood. In cerebral palsy spasticity is considered as a primary factor leads to much impairment which is inversely related to functional development that means greater the spasticity lowers the level of function. There are many ways to treat spasticity which involve stretching, strengthening, postural education, neuromuscular electrical stimulation, cryotherapy and myofascial release technique.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial. Study will be approved by ethical committee. After that informed consent will be taken and patients will be included in the study on the basis of inclusion criteria. Non probability convenience sampling technique will be used and study will be conducted on 28 patients with spastic hemiplegic cerebral palsy, 6 to 12 years of age. Patient will be randomly categorize into two groups by using flip coin. Experimental group will receive myofascial release on ankle planterflexors and quick icing treatment protocol on ankle dorsiflexors. Control group will receive only myofascial release treatment protocol on ankle planterflexors. Pre and Post intervention assessment will be made for both groups. Tone of planterflexors will be assessed by Modified Ashworth Scale, ankle passive range of motion will be assessed by goniometer and static balance will be assessed by Romberg test(open eyes).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with hemiplegic cerebral palsy
* Both genders
* Age between 6 to 12 years
* GMFCS Level I and II
* Modified Ashworth scale (grade1 - grade 3

Exclusion Criteria:

* Hypersensitive to cold
* Underwent any corrective surgery
* Specific perceptual and cognitive impairments
* Subjects who has received Botulinium toxin injection in the past 6 months

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 4 weeks
  Modified Ashworth Scale is a subjective 5-point scale. The modified Ashworth scale is the most universally accepted clinical tool used to measure the increase of muscle tone. The modified Ashworth scale is a muscle tone assessment scale used to assess the resistance experienced during passive range of motion, which does not require any instrumentation and is quick to perform. The MAS is the gold standard for the measurement of new assessment tools and has shown to have good intrarater reliability (0.84) and good interrater reliability(0.83).Modified Ashworth Scale is used as a qualitative scale in this study
Romberg test (open eyes) | 4 weeks
  The Romberg test is a simple bedside test that should be performed on all patients presenting with imbalance. In the Romberg test with eyes open, the patient is asked to remove shoes and stand with both feet together. Next, the examiner instructs the patient to hold their arms next to the body or crossed in front of the body. The test involves asking the patient to keep their eyes open while the examiner assesses the patient's body movement relative to balance. Romberg sign is positive if the patient is often unsteady with the eyes open
Goniometer | 4 weeks
  Goniometer is implemented as quantifiable monitoring device(9). For both upper and lower limb. It is the most extended tool for measuring ROM in the clinical practice. Goniometry is quantifiable monitoring device. Intertester and intratester believability towards goniometric measures at ankle joint are 0.86 and 0.90 in terms of ICC

CONTACTS AND LOCATIONS:
Overall Officials: Minal Fatima, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whisler SL, Lang DM, Armstrong M, Vickers J, Qualls C, Feldman JS. Effects of myofascial release and other advanced myofascial therapies on children with cerebral palsy: six case reports. Explore (NY). 2012 May-Jun;8(3):199-205. doi: 10.1016/j.explore.2012.02.003. No abstract available. PMID 22560759